CLINICAL TRIAL: NCT03389308
Title: An International, Multicenter, Open-label, Long Term Extension Study Evaluating the Safety of Diacerein 1% Ointment Topical Formulation in Subjects With Epidermolysis Bullosa Simplex (EBS)
Brief Title: Long Term Open-label Study Evaluating Safety of Diacerein 1% Ointment Topical Formulation in Subjects With Epidermolysis Bullosa Simplex
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Castle Creek Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCP-020-302
Record Dates: First submitted 2017-12-19; First posted 2018-01-03 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Epidermolysis Bullosa; Epidermolysis Bullosa Simplex
Keywords: Epidermolysis Bullosa (EB); Epidermolysis Bullosa Simplex (EBS)
MeSH Terms: conditions — Epidermolysis Bullosa; Epidermolysis Bullosa Simplex | interventions — diacerein; Ointments

STUDY DESIGN:
Intervention Model Description: This is an international, multicenter, open-label, long term extension study evaluating the safety of topical Diacerein 1% Ointment for the treatment of subjects with EBS. At Baseline Visit, EBS subjects who participated the CCP-020-301 double-blind safety and efficacy study or participated in the CCP-020-101 PK study (feeder studies) and who meet all the inclusion/exclusion criteria will be eligible to enroll in this study.
Masking Description: Each treatment cycle will consist of 8 weeks on treatment, followed by 8 weeks off treatment with a maximum of 2 treatment cycles allowed for up to 1 year. Subjects should be assessed at minimum every 8 weeks for disease activity. Once a subject completes two cycles of treatment or reaches Week 52, the subject will be discharged from the study. Subjects may not start a new treatment cycle past Week 36 from Baseline Visit without prior sponsor approval. The duration of a subject's participation in the extension study may be as short as 32 weeks or as long as 52 weeks depending on the cycle initiation schedule for each individual subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment period (Experimental): Subjects with active lesions as determined Investigator's clinical assessment, will initiate a cycle of applying diacerein 1% ointment once-daily, study medication, at home to their EBS lesions for 8 weeks.
  Following the Treatment Period, subjects will go Off Treatment for 8 weeks using only investigator approved bland, non-medicated emollient/moisturizer, routine cleansing products and sunscreens. As determined Investigator's clinical assessment, subjects may enter into another Treatment Period of 8 weeks.
  The duration of a subject's participation in the extension study may be as short as 32 weeks or as long as 52 weeks depending on the cycle initiation schedule for each individual subject.
  Interventions: Drug: diacerein 1% ointment

INTERVENTIONS:
Drug: diacerein 1% ointment — Topically apply study medication to lesions identified by the Investigator that require.
  treatment
  Other Names: CCP-020

SUMMARY:
The primary objective of this study is to evaluate the long term safety and tolerability of diacerein 1% ointment for 2 treatment cycles in subjects with EBS that previously participated in the CCP-020-301 or the CCP-020-101 studies.

DETAILED DESCRIPTION:
This is an international, multicenter, open-label, long term extension study evaluating the safety of topical Diacerein 1% Ointment for the treatment of subjects with EBS. At Visit 1, EBS subjects who completed the CCP-020-301 double-blind safety and efficacy study or participated in the CCP-020-101 PK study (feeder studies) who meet all the inclusion/exclusion criteria will be eligible to complete 2 treatment cycles of CCP-020.

Each treatment cycle will consist of 8 weeks on treatment (once-daily, at home study medication applications) followed by 8 weeks off treatment (only Investigator approved bland, non-medicated emollient/moisturizer, routine cleansing products and sunscreens) with a maximum of 2 treatment cycles allowed for up to 52 weeks.

At Baseline Visit (corresponding to the final study visit of the feeder study), the investigator will perform a clinical assessment and determine if any of the subject's lesions require treatment (up to 30% BSA). If the subject has active lesions as determined by the Investigator's clinical assessment, the subject will initiate a cycle of once-daily, at home study medication application to their EBS lesions for 8 weeks (treatment period) followed by an 8-week period where no treatment will be administered. Subjects presenting with no active lesions (as determined by the Investigator's clinical assessment) will not begin treatment and instead, will be instructed to return to the clinic for re-evaluation in 8 weeks or upon worsening of EBS lesions, whichever happens first.

ELIGIBILITY:
Key Inclusion Criteria:

* The subject is capable of understanding and complying with protocol requirements.
* The subject or the subject's legally acceptable representative signs and dates a written, informed consent/assent form and any required privacy authorization prior to the initiation of any study procedures.
* Subject has a documented genetic mutation consistent with EBS.
* Subject has completed study CCP-020-301 or participated in study CCP-020-101.
* Subject/caregiver agrees to report use of any topical therapies applied to EBS lesions
* If the subject is a woman of childbearing potential, she has a negative urine pregnancy test and agrees to use an approved effective method of birth control, for the duration of the study.
* Subject is non-lactating and is not planning for pregnancy during the study period.
* Subject is willing and able to follow all study instructions and to attend all study visits.

Key Exclusion Criteria:

* Subject has EBS lesions to be treated that are infected
* Subject has evidence of a systemic infection or has used systemic antibiotics within 7 days prior to Baseline Visit.
* The subject was discontinued from the feeder study due to an adverse event judged to be related or possibly related to the study medication.
* Subject has experienced a change in clinical status from the feeder study that puts the subject at undue risk to participate.

Ages: 6 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Spellman, MD, Study Chair — Castle Creek Pharmaceuticals
Locations (3):
- United States (3):
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of North Carolina (UNC) - Chapel Hill, Chapel Hill, North Carolina
  - Children's Hospital of San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Diacerein 1% Ointment: Subjects with active lesions as determined Investigator's clinical assessment, will apply diacerein 1% ointment once-daily, to their EBS lesions for 8 weeks. Following an off treatment period of 8 weeks or more, subjects may enter into another Treatment Period of 8 weeks. The subject's participation may range from 32 weeks to 52 weeks.
Period: Overall Study
Arm/Group | Diacerein 1% Ointment
Started | 51
Completed | 39
Not Completed | 12
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 3
Not completed — Adverse Event | 2
Not completed — Sponsor Request | 2

BASELINE CHARACTERISTICS:
Arm/Group | Diacerein 1% Ointment
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.6 (10.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 1
  Israel | 5
  Australia | 2
  United Kingdom | 7
  Netherlands | 3
  France | 9
  Germany | 2
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events
Description: Number and percentage of participants with any treatment-emergent adverse event.
Time Frame: up to 52 weeks
Population: Safety population: All subjects who received at least one application of diacerein 1% ointment.
Measure: Count of Participants; unit: Participants
Arm/Group | Diacerein 1% Ointment
Number analyzed (Participants) | 51
Participants | 40

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Arm/Group | Diacerein 1% Ointment
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 21/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diacerein 1% Ointment (N=51)
Nasopharyngitis (Infections and infestations) | 7 (10)
Skin infection (Infections and infestations) | 5 (9)
Ear infection (Infections and infestations) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 3 (3)
Pyrexia (General disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT03389308/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT03389308/SAP_001.pdf